CLINICAL TRIAL: NCT02922634
Title: Preoperative Cognitive Screening in Older Spinal Surgical Patients: Feasibility and Utility for Predicting Morbidity
Brief Title: Preoperative Cognitive Screening in Older Spinal Surgical Patients
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Deborah Culley, MD, Dr., Brigham and Women's Hospital
Other Study IDs: 2016P000012
Record Dates: First submitted 2016-03-14; First posted 2016-10-04 (Estimated); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Cognitive Impairment; Frail Elderly Syndrome
Keywords: postoperative health outcomes; older surgical patients; delirium
MeSH Terms: conditions — Cognitive Dysfunction; Delirium | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- older surgical patients: Older surgical patients presenting for elective spine surgery
  Interventions: Other: Mini Cog

INTERVENTIONS:
Other: Mini Cog — short cognitive screen, short Frailty screen
  Other Names: Frailty; Animal Fluency

SUMMARY:
The objectives of this study are to determine whether identifying patients with baseline cognitive deficits or frailty predict postoperative delirium.

DETAILED DESCRIPTION:
This project is designed as a prospective, single-center observational study. The cohort will consist of 229 consenting subjects ≥ 70 years of age who present to the Brigham and Women's Hospital Weiner Center for Preoperative Evaluation (CPE) prior to elective spine surgery. These ages are chosen as significant clinical data demonstrate increased cognitive impairment in community dwelling elders. Eligibility criteria include: patients ≥ 70 years of age with an American Society of Anesthesiologists (ASA) physical status classification of I-III presenting for elective spine surgery. Exclusion criteria will include planned Intensive Care Unit (ICU) admission postoperatively, history of stroke or brain tumor, uncorrected vision or hearing impairment (unable to see pictures or read or hear instructions); limited use of the dominant hand (limited ability to draw); and or inability to speak, read, or understand English.

Patients will be introduced to the study through a flyer provided to them in their surgeon's office. A study team member will speak with those favorably predisposed to participate to determine if they satisfy eligibility criteria. After obtaining consent, study staff will gain information about the patient's age and years of education. Study staff will administer Health and functional status activities of daily living (ADLs) and instrumental activities of daily living (IADLs), respectively, and the World Health Organization Disability Assessment Scale [WHODAS]) will be administered to all surgical patients. The World Health Organization Disability Assessment Schedule 2.0 is an alternative to the 36-Item Rand Health Survey Short-Form (SF36) to measure physical health and disability. In addition, all patients will be asked if they've had a fall within the last 6 months, whether they've been evaluated for a change in memory or thinking, who accompanied them to their appointment, their employment status and their living situation (alone, institutionalized, living with family members) in a patient survey. The study staff will administer the MiniCog, a simple cognitive screening tool that takes just 2-4 min to complete and has little or no education, language, or race bias. In addition, the Animal Fluency test will be administered, which is a short cognitive screen that takes one minute to complete. Frailty will be measured using the Frail Scale. Other measures of cognitive impairment will be obtained by study staff through: documentation on the patient's standard preoperative form, patient or informant report of diagnosis or evaluation for cognitive impairment or memory concerns, and systematic medical record review. Each enrolled patient will receive a business card listing the investigators' contact information and be advised to expect a follow up telephone up to 6 and 12 months after surgery to verify data elements and reassess functional outcome.

Delirium will be assessed prospectively once per day on postoperative days 1, 2, and 3 if the patient remains hospitalized, by a trained study team member using the Confusion Assessment Method [CAM]. For patients that are in the Intensive Care Unit (ICU) postoperatively, the Confusion Assessment Method for the ICU (CAM-ICU) will be administered prospectively twice per day on postoperative days 1, 2, and 3 if the patient remains hospitalized by a trained study team member (Attachment-CAM-ICU). Delirium is most common on postoperative days 1-3 and the CAM is a well-validated measure of delirium in surgical patients. For functional status, the WHODAS will be administered 6-12 months postoperatively either by personnel in the surgeon's office as part of routine follow up or by study staff or by telephone. We will also collect information on secondary outcomes including discharge to place other than home (rehabilitation, skilled nursing facility), hospital length of stay (LOS), 30-day reoperation or readmission rate, and 30-day mortality. These outcomes are recorded in the medical record, the BWH Balanced Scorecard, an electronic database of all hospitalized patients that tabulates 31 elements of the hospital event, or the Brigham and Women's Hospital BWH Research Patient Database Enhanced Query. Data will also be confirmed by a follow up telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* patients 70 years of age and older presenting to the BWH Weiner Center for Preoperative Evaluation
* undergoing elective spine surgery

Exclusion Criteria:

* include planned ICU admission postoperatively
* history of stroke or brain tumor
* uncorrected vision or hearing impairment (unable to see pictures or read or hear instructions)
* limited use of the dominant hand (limited ability to draw)
* inability to speak, read, or understand English.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 229 consenting subjects ≥ 70 years of age who present to the BWH Weiner Center for Preoperative Evaluation (CPE) prior to elective spine surgery.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2019-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Culley, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Weiner Center for Preoperative Evaluation, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 17, 2017 and October 9, 2018, study staff members recruited patients ≥ 70 yr of age scheduled for elective spine surgery at the Brigham and Women's Hospital and were expected to have an inpatient admission after their procedure. We selected this patient population because spine surgery is the third most common surgical procedure in older persons18 and our previous work showed that nearly 20% of this surgical demographic develops delirium postoperatively.
Pre-assignment Details: Older patients ≥ 70 years of age presenting for elective spine surgery.
Groups:
- Older Surgical Patients Having Spine Surgery: Older surgical patients (≥ 70 years of age) presenting for elective spine surgery.
Period: Overall Study
Arm/Group | Older Surgical Patients Having Spine Surgery
Started | 229
Completed | 219
Not Completed | 10
Not completed — Withdrawal by Subject | 5
Not completed — Did not have their surgery | 5

BASELINE CHARACTERISTICS:
Population: Patients ≥ 70 yr of age who were scheduled for elective spine surgery expected to have an inpatient admission after their procedure. Patients were identified in the preoperative evaluation schedule in the electronic medical record. 5 of these patients withdrew from the study and 5 did not have their surgical procedure thus 219 patients were analyzed.
Groups:
- Older Surgical Patients: Older surgical patients presenting for elective spine surgery by neurosurgeons Dr. Groff, Dr. Lu and Dr. Chi
  Mini Cog: short cognitive screen, short Frailty screen
Arm/Group | Older Surgical Patients
Number analyzed (Participants) | 219
Age, Categorical [Count of Participants; unit: Participants] — Population: 5 patients withdrew from the study, 5 patients did not have their surgery
  Participants
    <=18 years | 0
    Between 18 and 65 years | 0
    >=65 years | 219
Age, Continuous [Median (Inter-Quartile Range); unit: Year] — collected from the medical record Population: 5 Patients withdrew from the study, 5 patients did not have surgery
  Year | 75 [73 to 79]
Sex: Female, Male [Count of Participants; unit: Participants] — binary sex, male or female Population: 5 patients withdrew from the study and 5 patients did not have surgery
  Participants
    Female | 95
    Male | 124
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 219
Frail Scale [Count of Participants; unit: Participants] — 5 point scale with score of 0 meaning robust, 1-2 pre-frail, and scores of 3-5 frail. Population: 5 patients withdrew from the study, 5 patients did not have their surgery and 1 patient left before completing the frail scale.
  Participants
    number analyzed (Participants) | 218
    Score 0 | 48
    Score 1-2 | 117
    Score 3-5 | 53
Mini-Cog [Median (Inter-Quartile Range); unit: units on a scale] — The Mini-Cog is a brief cognitive screening test for visuospatial representation, recall, and executive function. The test involves that includes recalling three words (banana, sunrise, and chair) and a clock drawing. The Mini-Cog has a scale from 0 to 5, and a score of ≥ 3 indicates better cognitive outcomes. One point is designated for each of 3 words recalled and up to two points for the clock drawing component. Population: 5 patients withdrew from the study and 5 patients did not have surgery
  units on a scale | 4 [3 to 5]
Animal Verbal Fluency [Mean (Standard Deviation); unit: animals] — Number of unique animals the patient can say in 1 minute. Higher number of animals named in 1 minute reflects better cognitive performance Population: 5 patients withdrew from the study and 5 patients did not have surgery
  animals | 18 (6)
Surgical Invasiveness [Count of Participants; unit: Participants] — Surgical invasiveness on a 4 point scale. The stages were categorized clinically as the following: Tier 1 for microdiscectomy, Tier 2 for lumbar laminectomy, anterior cervical, minimally invasive, foraminotomy, facetectomy, Tier 3 for lumbar fusion, trauma, and post-cervical, and Tier 4 for tumor, infection, deformity, and anterior and posterior cervical. Higher tiers indicate greater levels of invasiveness. Since there were very few patients with an invasiveness of 1 or 4 they were placed into two groups, with invasiveness levels I and 2 or 3 and 4. Population: 5 patients withdrew from the study and 5 patients did not have their surgery
  Participants
    Tier 1 and 2 | 111
    Tier 3 and 4 | 108
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] — Population: 5 of these patients withdrew from the study and 5 did not have their surgical procedure and 2 patients did not have their BMI recorded in the medical record
  kg/m^2
    number analyzed (Participants) | 217
    (all) | 28 [25 to 32]
Level of education [Count of Participants; unit: Participants] — Patients were divided into those that had less than a bachelors degree, and those that had a bachelors degree or higher Population: 5 of these patients withdrew from the study and 5 did not have their surgical procedure. An additional 7 did not provide information on their level of education.
  Participants
    number analyzed (Participants) | 212
    Bachelors degree or higher | 144
    Less than a bachelors degree | 68
ASA Physical Status [Count of Participants; unit: Participants] — Scaled score with lower scores having a better functional status than a higher score. Population: 5 patients withdrew from the study and 5 patients did not have their surgery.
  Participants
    ASA 1 or 2 | 70
    ASA 3 or 4 | 149
Metabolic equivalents of task [Count of Participants; unit: Participants] — scaled score where a higher number means the patient is more physically fit. Population: 5 of these patients withdrew from the study and 5 did not have their surgical procedure and an additional 10 patients did not have this noted in their medical record.
  Participants
    number analyzed (Participants) | 209
    METS < 4 | 60
    METS ≥ 4 | 149
Total number of medications [Median (Inter-Quartile Range); unit: total number of medications] — Population: 5 patients withdrew from the study and 5 patients did not have their surgery
  total number of medications | 8 [5 to 11]
Preoperative use of opioids [Count of Participants; unit: Participants] — Population: 5 patients withdrew from the study and 5 patients did not have their surgery
  Participants
    preoperative opioid use | 55
    No preoperative use of opioids | 164
Alcohol consumption [Count of Participants; unit: Participants] — patient consumed alcohol preoperatively Population: 5 patients withdrew from the study and 5 patients did not have their surgery.
  Participants
    Yes | 125
    No | 94
History of depression [Count of Participants; unit: Participants] — Population: 5 patients withdrew from the study and 5 patients did not have their surgery
  Participants
    Yes | 39
    No | 180
Psychiatric History [Count of Participants; unit: Participants] — History of psychiatric illness Population: 5 patients withdrew from the study and 5 patients did not have their surgery
  Participants
    Yes | 22
    No | 197

OUTCOME MEASURES:

1. Primary Outcome: Delirium by Age
Description: The median ages of patients who did or did not develop post-operative delirium as assessed by the Confusion Assessment Method. The Confusion Assessment Method (CAM) is a short diagnostic interview for CAM-defined delirium. Delirium is defined as the sudden change in someone's thinking ability that can have devastating consequences and can be very easily missed due to its frequent subtlety. The 4 CAM features assessed by the CAM include: acute onset or fluctuation, inattention, disorganized thinking, or altered level of consciousness.
Time Frame: up to 3 days post-op
Population: Patients over the age of 70 undergoing spinal surgeries
Measure: Median (Inter-Quartile Range); unit: years
Groups:
- No Delirium: Older surgical patients presenting for elective spine surgery that did not develop post-op delirium
- Delirium: Older surgical patients presenting for elective spine surgery that did develop post-op delirium
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
years | 75 [73 to 79] | 77 [72 to 80]
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.508, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Number of Participants With or Without Delirium by Sex
Description: Sex of patients who did or did not develop post-operative delirium as assessed by the Confusion Assessment Method.
Time Frame: up to 3 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
Participants
  Male | 94 | 30
  Female | 70 | 25
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.720, Chi-squared — The chi-squared test for both males and females with and without delirium

3. Primary Outcome: Delirium by Body Mass Index
Description: Median body mass index of patients who did or did not develop post-operative delirium as assessed by the Confusion Assessment Method.
Time Frame: up to 3 days post-op
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
kg/m^2 | 28 [25 to 32] | 30 [26 to 34]
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.025, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Number of Participants With or Without Delirium by College Degree
Description: Counts of patients with a college degree who did or did not develop post-operative delirium as assessed by the Confusion Assessment Method.
Time Frame: up to 3 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
Participants | 108 | 36
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.480, Chi-squared

5. Primary Outcome: Participants With an ASA Physical Status Score and the Development of Postoperative Delirium
Description: The ASA Physical Status Classification System assesses and communicates a patient's pre-anesthesia medical co-morbidities and is on a scale of I-VI. This study recruited patients with an ASA physical status of I-III. ASA I is defined as a normal healthy patient, ASA II is defined as a patient with a mild systemic disease, ASA III is defined as a patient with severe systemic disease. ASA physical status of patients who did or did not develop post-operative delirium as assessed by the Confusion Assessment Method.
Time Frame: up to 3 days post-op
Measure: Count of Participants; unit: Participants
Groups:
- No Delirium: Older surgical patients presenting for elective spine surgery with an ASA Physical that did not develop post-op delirium
- Delirium: Older surgical patients presenting for elective spine surgery with an ASA physical status of that did develop post-op delirium
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
Participants
  ASA Physical status of greater than or equal to 3 | 105 | 44
  ASA Physical Status of less than 3 | 59 | 11
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.028, Chi-squared

6. Primary Outcome: Number of Participants With or Without Delirium by Metabolic Equivalent of Task Score < 4
Description: Patients with a metabolic equivalent of task (METS) score < 4 who did or did not develop post-operative delirium as assessed by the Confusion Assessment Method. The METS score is a ratio of the working metabolic rate relative to the resting metabolic rate and is one way to describe the intensity of an exercise or activity. This was assessed by the preoperative or surgical study staff. A score of < 3 is for light intesity activities, 3-6 for moderate intensity activities, and ≥ 6 for vigorous intensity activities.
Time Frame: up to 3 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
Participants | 45 | 25
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.007, Chi-squared

7. Primary Outcome: Delirium by Total Number of Medications Taken at Baseline
Description: Median total number of medications of patients who did or did not develop post-operative delirium as assessed by the Confusion Assessment Method.
Time Frame: up to 3 days post-op
Measure: Median (Inter-Quartile Range); unit: medications
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
medications | 8 [5 to 10] | 9 [7 to 12]
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Number of Participants With or Without Delirium by Opioid Use
Description: Patients with chronic use of opioids who did or did not develop post-operative delirium as assessed by the Confusion Assessment Method.
Time Frame: up to 3 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
Participants | 34 | 21
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.01, Chi-squared

9. Primary Outcome: Number of Participants With or Without Delirium by Alcohol Consumption
Description: Patients who did or did not develop post-operative delirium as assessed by the Confusion Assessment Method based on alcohol consumption.
Time Frame: up to 3 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
Participants | 98 | 27
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.101, Chi-squared

10. Primary Outcome: Number of Participants With or Without Delirium by Presence of Depression
Description: Patients with depression who did or did not develop post-operative delirium as assessed by the Confusion Assessment Method.
Time Frame: up to 3 days post-op
Measure: Count of Participants; unit: Participants
Groups:
- No Delirium: Older spine surgery patients who did not develop post-operative delirium
- Delirium: Older spine surgery patients who did develop post-operative delirium
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
Participants | 26 | 13
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.192, Chi-squared

11. Primary Outcome: Number of Participants With or Without Delirium by Psychiatric History
Description: Patients with a history of psychiatric disorders who did or did not develop post-operative delirium as assessed by the confusion assessment method.
Time Frame: up to 3 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
Participants | 14 | 8
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.200, Chi-squared

12. Primary Outcome: Delirium by Mini-cog Score
Description: Median mini-cog score of patients who did or did not develop post-operative delirium as assessed by the confusion assessment method. The Mini-Cog is a brief cognitive screening test for visuospatial representation, recall, and executive function. The test involves that includes recalling three words (banana, sunrise, and chair) and a clock drawing. The Mini-Cog has a scale from 0 to 5, a with higher scores suggesting better cognitive performance. One point is designated for each of 3 words recalled and up to two points for the clock drawing component.
Time Frame: up to 3 days post-op
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
scores on a scale | 4 [3 to 5] | 4 [2 to 5]
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.333, Wilcoxon (Mann-Whitney)

13. Primary Outcome: Number of Participants With or Without Delirium by FRAIL Score
Description: Robust, pre-frail, and frail patients who did or did not develop post-operative delirium as assessed by the confusion assessment method.
Time Frame: up to 3 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 54
Participants
  Robust (score 0) | 43 | 5
  Pre-frail (score 1 and 2) | 92 | 25
  Frail (score 3-5) | 29 | 24
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.001, Chi-squared — This is a chi-squared test between the FRAIL categories for participants with or without delirium

14. Primary Outcome: Number of Participants With or Without Delirium by Surgical Invasivness
Description: Surgical invasiveness for patients who did or did not develop post-operative delirium as assessed by the confusion assessment method. The levels of invasiveness were categorized clinically as the following: Tier 1 for microdiscectomy, Tier 2 for lumbar laminectomy, anterior cervical, minimally invasive, foraminotomy, facetectomy, Tier 3 for lumbar fusion, trauma, and post-cervical, and Tier 4 for tumor, infection, deformity, and anterior and posterior cervical. Higher tiers indicate greater levels of invasiveness. Since there were very few patients with an invasiveness of 1 or 4 they were placed into two groups, with invasiveness levels I and 2 or 3 and 4.
Time Frame: up to 3 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | No Delirium | Delirium
Number analyzed (Participants) | 164 | 55
Participants
  Tier 1 + 2 | 93 | 18
  Tier 3 + 4 | 71 | 37
Statistical Analysis 1: Comparison: No Delirium vs Delirium; Test type: Superiority; p = 0.002, Chi-squared — This is a chi-squared test of the categories for levels of invasiveness for participants with or without delirium

15. Secondary Outcome: Number of Participants With In-hospital Complications Were Observed During Their Length of Stay in the Hospital With Death Postoperative Death Monitored up to Day 30.
Description: In hospital complications after the surgical procedure including: Myocardial Infarction, congestive heart failure (CHF), Cardiac Arrest, Arrythmia, Pneumonia, pulmonary embolism (PE), Reintubation, Stroke, Delirium, Coma>24h, deep wound infection,Superficial wound infection, Sepsis, Renal Failure, urinary tract infection (UTI), Reoperation, deep vein thrombosis (DVT), intensive care unit (ICU) admission,
Time Frame: duration of hospital stay, up to 30 days
Population: All spine surgery patients enrolled in the study.
Measure: Count of Participants; unit: Participants
Groups:
- In Hospital Complications: Patients that experienced in hospital complications not including post-operative delirium.
Arm/Group | In Hospital Complications
Number analyzed (Participants) | 219
Participants
  no in-hospital complications | 151
  in-hospital complications | 68

16. Secondary Outcome: Participants' Discharge Location (Home vs. Other Than Home)
Description: Location where patients were discharged (Home vs other than home) on the day of patients discharge from the hospital.
Time Frame: up to 30 days after the surgical procedure
Measure: Count of Participants; unit: Participants
Groups:
- Discharge Location: Discharge location (home vs place other than home) for patients who participated in this study.
Arm/Group | Discharge Location
Number analyzed (Participants) | 219
Participants
  Home | 138
  Place other than home | 77
  Not documented | 4

ADVERSE EVENTS:
Time Frame: The patients were observed for postoperative complications during their hospital length of stay and death monitored up to postoperative day 30
Description: This was an observational study that only followed patients through their length of stay in the hospital with the exception of 30 day mortality. No patients were identified with 30 day mortality
Groups:
- Postoperative Outcomes in Older Patients After Spine Surgery: Older surgical patients that had elective spine surgery and developed an in-hospital cardiopulmonary, infectious, renal or cerebrovascular complication.
Arm/Group | Postoperative Outcomes in Older Patients After Spine Surgery
All-Cause Mortality (participants affected / at risk) | 0/219
Serious Adverse Events (participants affected / at risk) | 0/219
Other Adverse Events (participants affected / at risk) | 0/219

LIMITATIONS AND CAVEATS:
Thirty percent of eligible patients declined participation in this study leading to potential selection bias based on the type of person who chooses to participate in such a study. There is also the possibility that we underestimated the prevalence of post-operative delirium because we only assessed patients for delirium once a day for 3 days post-op and by systematic chart review.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT02922634/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT02922634/ICF_001.pdf